CLINICAL TRIAL: NCT04455672
Title: A Comparative Study Using Two 3D Printed Occlusal Splints for Patients With Tempromandibular Disorder (A Randomized Cross Over Clinical Trial)
Brief Title: A Comparative Study Using Two 3D Printed Occlusal Splints for Patients With Tempromandibular Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mostafa mohamed sobhy, the principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEBD-CU-2020-06-29
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Temporomandibular Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Splints

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional group (Experimental): patient using two types of splints (3d Anterior Rrepositioning Splint then printed stabilizing splint)
  Interventions: Device: splints
- control group (Active Comparator): patient using two types of splints (3d printed stabilizing splint then Anterior Rrepositioning Splint)
  Interventions: Device: splints

INTERVENTIONS:
Device: splints — * Scaning of the maxillary and mandibular cast in the centric relation.
  * The CAD/ CAM splints will be designed using Exocad s.
  * The design will include all maxillary teeth and the occlusal surfaces will be flat and smooth.
  * The difference in design between the ARS and the stabilization splint, is that the ARS will have an anterior ramp to allow for posterior disocclusion of posterior teeth, while the stabilization splint will not have such a pronounced anterior ramp.
  * Both splints will be printed using Dent2 3D printer and then cured using Dentcure.
  * All patient will be asked to wear their spints during sleeping only.
  * In each group, patient will be recalled after 1week,2 weeks 1,2and 3monthes then change for the other splint for another 3 months .

SUMMARY:
• to compare the relief of pain for patients with anterior disc displacement with reduction between two groups; in the first group a digitally formed stabilizing splint followed by an anterior repositioning splint (ARS) and the second group a digitally fabricated (ARS) splints followed by a stabilizing splints

ELIGIBILITY:
Inclusion Criteria:

* • TMDs according to the research diagnostic criteria (RDC)8 which include: i. Painful TMJ audible and palpable click unilateral or bilateral ii. Presence of clicking during opening. iii. TMJ tenderness.

  * Fully dentate patients without any malocclusion (natural or restored by fixed prothesis) and good oral hygiene.
  * Co-operative patient that should show motivation to follow up.

Exclusion Criteria:

* • Patients with systemic diseases which could affect TMJ, e.g., rheumatoid arthritis, osteoarthrosis, Myasthenia Gravis and fibromyalgia.

  * Patients taking analgesic, muscle relaxant, or anti-inflammatory drugs were excluded because such drugs could influence the results.
  * Patients with removable dental prosthesis

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-07-26 (Estimated); Study Completion 2021-09-26 (Estimated)

PRIMARY OUTCOMES:
pain relief | 6 months
  questionnaire will be used to evaluate the pain